CLINICAL TRIAL: NCT06997289
Title: Intelligent Complementary Diagnosis and Treatment of Traditional Chinese Medicine for Primary Insomnia
Brief Title: Intelligent Approach to Traditional Chinese Medicine for Insomnia
Acronym: TCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-10-005C
Record Dates: First submitted 2025-02-10; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Insomnia
Keywords: auricular points,; Chinese medicine; pulse diagnosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Randomized controlled cross-over experimental design (Experimental): Struggling to fall asleep or stay asleep, experiencing frequent awakenings, or finding it challenging to return to sleep after waking up.
  Waking up early in the morning and being unable to go back to sleep. Sleep disturbances leading to significant distress or impairment in various aspects of life such as social, occupational, or academic functioning.
  Experiencing difficulty sleeping on at least three nights a week for a period of at least three months.
  No use of hypnotic or stable use of hypnotic and no medication adjustment in the past month
  Interventions: Drug: Group that is receiving treatment.

INTERVENTIONS:
Drug: Group that is receiving treatment. — Incorporate the following regimen into your daily routine for optimal health benefits:
  Chinese Medicine: Take a combination of Modified Xiaoyao Powder (2g), Tianwang Buxin Dan (1.5g), Wendan Decoction (0.5g), Night Jiaoteng (0.5g), and Fushen (0.5g) twice a day for a duration of 1 month. This regimen comes from Keda GMP Pharmaceutical Factory.
  Auricular Point Stimulation: Apply small 0.2cm ear magnetic beads on the Shenmen, heart, and brainstem points on both sides of the ear.
  Consistency is key to achieving positive results, so make sure to follow this routine diligently.
  Two treatment methods are carried out simultaneously
  Other Names: Auricular acupuncture

SUMMARY:
Insomnia is a very common health issue, affecting over 40% of the population in Chinese-speaking regions. The impact of insomnia on society, economy, mental health, and physical health is significant, with previous research indicating that insomnia is associated with an increased risk of high blood pressure, heart disease, anxiety, and depression, which can ultimately lead to a decline in quality of life. Treatment for insomnia includes non-pharmacological and pharmacological interventions, with clinical practice often utilizing sedative medications for sleep, but with side effects such as dependency, tolerance, daytime drowsiness, and withdrawal symptoms, which make it challenging for patients to find suitable medical treatment. Traditional Chinese Medicine (TCM) approaches insomnia by first conducting a thorough assessment based on individualized patterns (differentiation of body constitution) and evaluating insomnia-related symptoms, followed by an examination of tongue and pulse to determine the correct treatment plan, which may involve acupuncture, herbal medicine or a combination of both (integrative treatment). Due to the complex nature of insomnia, a definitive diagnosis requires neuroimaging and other measures during sleep studies to assess brain wave activity, if possible, to understand the cognitive impact.

DETAILED DESCRIPTION:
In the treatment of insomnia, Chinese medicine first assesses the individual's constitution and symptoms related to insomnia, before incorporating auricular acupuncture and pulse diagnosis. Subsequently, different syndrome types are identified and treated with acupuncture or traditional Chinese medicine (dialectical treatment). Since insomnia is often subjective, a definitive diagnosis may require overnight monitoring of brain waves and other parameters in a sleep laboratory. Smart imaging methods can help detect special reaction areas of ear points, while pulse diagnosis equipment can provide objective auxiliary diagnosis and classification of insomnia through pulse wave digital conversion analysis. Previous studies have demonstrated the effectiveness of auricular point stimulation in treating insomnia, and this study aims to enhance the therapeutic outcomes for primary insomnia by combining Chinese medicine techniques.

ELIGIBILITY:
Inclusion Criteria:

* Major mental illnesses include schizophrenia, bipolar disorder, major depression, dementia, apnea, restless legs syndrome, alcohol and substance abuse, organic psychosis and those with major physiological illnesses that affect sleep.

Exclusion Criteria:

* As per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) published by the American Psychiatric Association, insomnia is characterized.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire evaluation | up to 4 weeks"
  Pittsburgh Sleep Quality Index, PSQI)